CLINICAL TRIAL: NCT03069651
Title: A Prospective Randomised Pilot Study of Videoconferencing in Adults With Cystic Fibrosis Receiving Intravenous Antibiotics for Acute Pulmonary Exacerbations (VIRTUALCF)
Brief Title: Virtual Care in CF (VIRTUAL-CF) Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Heart of England NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2014134RM
Record Dates: First submitted 2016-12-09; First posted 2017-03-03 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — Telemedicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Virtual Care (Active Comparator): Subjects randomly allocated to receive 'virtual care' will be shown how to use the oximeter and spirometer, as well as the videoconferencing software.
  'Virtual care' subjects will be asked to perform a lung function test (using the spirometer) and record their oxygen saturations (using the oximeter) twice weekly during the videoconference with the CF team.
  Interventions: Other: Virtual Care
- Routine Care (Placebo Comparator): Usual clinical care.
  Interventions: Other: Virtual Care

INTERVENTIONS:
Other: Virtual Care — The use of Videoconferencing software to enable remote access to monitor patients in the 'Virtual Care' cohort.

SUMMARY:
Cystic fibrosis (CF) is the most common fatal inherited condition in Caucasians, causing recurrent chest infections (pulmonary exacerbations). People with CF experiencing pulmonary exacerbation often require a 14day course of intravenous antibiotics and this treatment can either be delivered in hospital or in the community. Patients admitted to hospital are seen regularly by members of the CF multidisciplinary team (MDT), including doctors, nurses, dieticians and physiotherapists. This allows patients' progress to be closely monitored and also gives patients the opportunity to discuss any concerns or questions. In contrast, patients receiving IV antibiotics in the community are only seen by the MDT at the beginning and end of their 14 day course of IV antibiotics. Although CF nurses often visit patients on 12 occasions during the course of treatment, patients are not routinely reassessed by the rest of the MDT. There is therefore less opportunity for the MDT to adjust patients' treatment and for patients to communicate with the MDT.

We therefore aim to study whether patients receiving IV antibiotics in the community benefit from monitoring their own oxygen saturations and lung function, as well as taking part in twice-weekly videoconferences with the MDT ('virtual care'). We expect that this will enable the MDT to to assess patients' progress more closely and allow patients to communicate with the MDT more easily. We will assess whether this improves patients' experience of their care and whether this translates into improvements in health and economic outcomes.

One hundred subjects will be recruited over a 12month period, with 50 subjects allocated to 'virtual care' and 50 subjects allocated to 'routine care'. Subjects receiving 'routine care' will receive usual clinical care.

The research team are well placed to perform the study because we are part of a large CF centre with an excellent record in clinical research.

DETAILED DESCRIPTION:
Study design Subjects will be recruited and randomly allocated in a 1:1 ratio, by means of sealed envelopes, to receive either 'virtual care' or 'routine care' for the 14day course of communitydeliveredIV antibiotics. Subjects randomly allocated to receive 'virtual care' will be shown how to use the oximeter and spirometer, as well as the videoconferencing software.

'Virtual care' subjects will be asked to perform a lung function test (using the spirometer) and record their oxygen saturations (using the oximeter) twice weekly during the videoconference with the CF team. Times and dates for the videoconference will be arranged at a time that is convenient for the patient. Subjects will be able to videoconference using any internetenabled device (laptop, tablet, mobile phone) available for the patient's use, but this device will not be provided as part of the study. The videoconferencing software used for this study is Webex, which is widely used within the NHS for videoconferencing with patients and all data is fully encrypted. Subjects in both groups ('virtual care' and 'routine care') will be offered home visits by a CF nurse if required as usual and an appointment made in the outpatient clinic immediately after the course of intravenous antibiotics finishes as usual.

Both cohorts ('virtual care' and 'routine care') will be asked to complete the CFQR(a validated disease-specific health related quality of life questionnaire) at the beginning and end of their course of IV antibiotics. Subjects in both groups will also be asked to complete a satisfaction questionnaire at the end of the course of antibiotics. Patients receiving 'virtual care' will be specifically asked about the ease of use of the oxygen saturation and spirometer equipment, as well as the videoconferencing system. Data regarding participants' lung function, nutritional status and medications will be recorded during each clinic visit for both cohorts. Subjects in both cohorts will also be asked to record any costs related to their care throughout the course of treatment (e.g. travel, parking). The researchers will record the costs associated with caring for each participant (such as cost of nursing visits and staff time) and the cost of conducting the study (e.g. cost of the oxygen saturation monitor, spirometer and videoconferencing equipment).

The primary outcome is health-related quality of life (measured by CFQR) in subjects receiving 'virtual care' compared to subjects receiving 'routine care'. Our null hypothesis is that there will be no significant difference in the CFQR in subjects receiving 'virtual care' compared to subjects receiving 'routine care'. Secondary outcomes are: patient satisfaction with care, days on intravenous antibiotics, lung function and weight in subjects receiving 'virtual care' compared to subjects receiving 'routine care'. A health economic analysis will be conducted to determine whether 'virtual care' is value for money both from an NHS and a patient perspective.

ELIGIBILITY:
Inclusion Criteria:

1. CF diagnosis confirmed by clinical characteristics, sweat test +/- genetic testing
2. Age over 18 years
3. Patient has been assessed by the clinical team to require a course of community-delivered intravenous antibiotics
4. Patients who give informed consent.

Exclusion Criteria:

1. Patients who are currently participating in another clinical trial (excluding observational studies)
2. Pneumothorax or lung surgery within the previous 3 months, eye surgery (e.g. cataract operation) in the previous 4 weeks, or any other factor that prevents measurement of spirometry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-03-29 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Does 'virtual care' affect health-related quality of life in CF adults receiving IV antibiotics? | 12 months
  Participants allocated to 'Virtual Care' will be asked to measure their oxygen saturations ( using the oximeter provided) and measure their lung function (using the spirometer provided) during the the twice-weekly video conferences with the CF MDT. Participants allocated to 'routine care will continue to receive standard care.

SECONDARY OUTCOMES:
Patient satisfaction with 'virtual care' compared to 'routine care' | 12 months
  Participant in both groups will be asked to complete a CF questionnaire at the beginning and end of their course of IV antibiotics and also complete a satisfaction questionnaire at the end of their IV antibiotic course
Changes in lung function in subjects receiving 'virtual care' compared to 'routine care' | 12 months
  Lung function for both groups will be monitored throughout their time in the study to see if the 'virtual care' has any impact.
Changes in weight in subjects receiving 'virtual care' compared to 'routine care' | 12 months
  Weight for both groups will be monitored throughout their time in the study to see if the 'virtual care' has any impact.
Health economic analysis of 'virtual care' compared to 'routine care' from a patient and NHS perspective. | 12 months
  The data from both groups will be analysed to see if the experience of the participants translates into health and economic outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Edward F Nash, MD, Principal Investigator — Consultant Physician
Locations (1):
- Birmingham Heartlands Hospital, Birmingham, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: No